CLINICAL TRIAL: NCT03057314
Title: Exploratory, Open Label Study to Improve Function and Welfare of Late-stage Cancer Subjects by Amorphous Calcium Carbonate (ACC) Treatment, Administered Orally and Concomitantly With Inhalation
Brief Title: Improving Function,Welfare of Late-stage Cancer Subjects by ACC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recreuitment
Sponsor: Amorphical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCS-ONCO-004
Record Dates: First submitted 2017-01-29; First posted 2017-02-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Solid Malignancies, With or Without Lung Metastases

STUDY DESIGN:
Intervention Model Description: OPEN LABEL SINGLE ARM STUDY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amorphous calcium carbonate (Experimental): The investigation product will include:
  1. ACC tablets, containing 200 mg elemental calcium
  2. 1% ACC (i.e. 0.3% calcium) + 5 mL Water for Injection, as a sterile suspension
  Interventions: Drug: Amorphous Calcium Carbonate

INTERVENTIONS:
Drug: Amorphous Calcium Carbonate — Subjects will be administered with:
  1. ACC tablets, containing 200 mg elemental calcium
  2. 1% ACC (i.e. 0.3% calcium) + 5 mL Water for Injection, as a sterile suspension
  Other Names: ACC

SUMMARY:
To improve the function and welfare of late stage solid cancer subjects by:

* enabling subjects to benefit from a potentially promising drug under development
* assessing initial evidence of improvement in Pain VAS score
* assessing initial improvement in Performance Status (PS)
* assessing initial improvement in oxygen saturation whenever it is feasible

DETAILED DESCRIPTION:
To improve the function and welfare of late stage solid cancer subjects by:

* enabling subjects to benefit from a potentially promising drug under development
* assessing initial evidence of improvement in Pain VAS score
* assessing initial improvement in Performance Status (PS)
* assessing improvement in oxygen saturation whenever it is feasible/ dyspnea measurement (Modified Borg Scale)

ELIGIBILITY:
Inclusion Criteria

1. Males and females, age >18 years
2. Signed the informed consent
3. Late Stage Histologically proven advanced solid tumours for which no standard curative therapy exist who failed or refused anti-cancer treatment
4. Subject should not have any illness or condition deemed by the physician to contra-indicate treatment with ACC or may interfere with the assessment of the therapy
5. Performance Status: ECOG 0-3/ Karnofsky performance status >50
6. Life Expectancy : about 2 months
7. Hormonal therapy is allowed if needed
8. Patient is on conservative treatment for relieving his symptoms
9. Subjects within normal range of serum-corrected albumin calcium (between 7.0-10.5 mg/dl)
10. Acceptable haematology and biochemistry variables:

    WBC ≥3000/mm3 Absolute Neutrophil count ≥ 1500 /mm3 Platelet Count ≥ 100,000/mm3 Hemoglobin ≥ 9 g/dL Bilirubin ≤ 1.5 x ULN ALT and AST ≤ 2.5 x ULN; for patients with hepatic metastases, ALT and AST ≤ 5 x ULN PT/PTT ≤ 1.5 ULN
11. Subjects should have sufficient Vitamin D levels upon study entry, which is defined as 25(OH)D serum level >20 ng/mL (50 nmol/L) according to a document composed by the Food and Nutrition Board of the Institute of Medicine, USA. If the subject is Vitamin D insufficient or deficient, then a loading dose of Vitamin D3 will be administered during subject's enrollment or during the study as follows:

    1. If the serum 25(OH)D level is 12-20 ng/mL (30-50 nmol/L) then a loading oral dose of 50,000 IU of Vitamin D3 should be administered twice with 3-5 days in between the doses.
    2. If the serum 25(OH)D level is ≤ 12 ng/mL (30 nmol/L), then a loading oral dose of 50,000 IU of Vitamin D3 will be administered three times with 3-5 days in between the doses. Serum 25(OH)D levels will be checked 1-2 weeks following the last loading.

    Nevertheless, if levels of vitamin D levels will not be within the normal range after adjustment efforts, patients will not excluded from the study.
12. Regardless of Vitamin D levels, all subjects will receive a daily maintenance dose of 1000 IU Vitamin D3, which should be taken in the morning with breakfast.
13. Subjects receiving Denosumab or bisphosphonates are eligible. Denosumab or bisphosphonates can be administered during the study to alleviate bone metastasis pain.
14. Negative Pregnancy Test.

Exclusion Criteria:

1. Concurrent treatment with acute anti-cancer therapy
2. Hypercalcemia (serum calcium concentration > 12.0 mg/dL)
3. Clinical Significant Cardiovascular Disease
4. Known alcohol or drug abuse
5. Any psychiatric condition that would prohibit understanding or rendering of Informed Consent
6. Active Participation in Clinical Trial in the last 2 weeks prior to inclusion
7. Brain metastases or spinal cord compression unless asymptomatic or treated and stable off steroids and anti-convulsants for at least 1 month prior to study treatment.
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Assessing a change in Pain Visual Analog Score (VAS score) | Baseline and on weeks 0,1,2,3,4,5,8 and on week 11
  Visual Analog scale ranging from 0 up to 10 meaning that ; 0 = no pain(min) 10=unbearable pain(max)

SECONDARY OUTCOMES:
Assessing a change in Performance Status (PS): ECOG scale | Baseline and on weeks 0,1,2,3,4,5,8 and on week 11
  assessing the patients improvement or not in their performance status;0 Fully active, able to carry on all pre-disease performance without restriction.1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.2 Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.3 Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair.5 Dead

CONTACTS AND LOCATIONS:
Overall Officials: Julia Rothman, Dr., Study Director — Head of clinical affairs
Locations (1):
- Meir, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No